CLINICAL TRIAL: NCT01949532
Title: An Open-Label, Single Arm, Phase 1 Study of the Pharmacokinetics and Safety of Carfilzomib in Subjects With Relapsed Multiple Myeloma and End-stage Renal Disease
Brief Title: Study of the Pharmacokinetics and Safety of Carfilzomib in Patients With Multiple Myeloma and Renal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CFZ001; 20130401 (Other: Sponsor)
Record Dates: First submitted 2013-09-06; First posted 2013-09-24 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Relapsed Multiple Myeloma; End-stage Renal Disease
MeSH Terms: conditions — Multiple Myeloma; Kidney Failure, Chronic | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Renal Function (Experimental): Participants with normal renal function (creatinine clearance [CrCl] ≥ 75 mL/min) received carfilzomib 20 mg/m² intravenous infusion (IV) on days 1 and 2 of cycle 1, followed by 27 mg/m² IV on days 8, 9, 15, and 16 of cycle 1. Participants who adequately tolerated dosing at 27 mg/m² received carfilzomib 56 mg/m² IV on days 1, 2, 8, 9, 15 and 16 of cycle 2 and all subsequent cycles. Participants continued treatment until confirmed progressive disease, unacceptable toxicity, withdrawal of consent, study closure, or death.
  Interventions: Drug: Carfilzomib
- End Stage Renal Disease (Experimental): Participants with end-stage renal disease (on hemodialysis) received carfilzomib 20 mg/m² intravenous infusion (IV) on days 1 and 2 of cycle 1, followed by 27 mg/m² IV on days 8, 9, 15, and 16 of cycle 1. Participants who adequately tolerated dosing at 27 mg/m² received carfilzomib 56 mg/m² IV on days 1, 2, 8, 9, 15 and 16 of cycle 2 and all subsequent cycles. Participants continued treatment until confirmed progressive disease, unacceptable toxicity, withdrawal of consent, study closure, or death.
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib was administered by IV injection.
  Other Names: Kyprolis®

SUMMARY:
The purpose of this study is to see how the body and the cancer react to carfilzomib, including measuring the amount of the study drug in the blood at certain times following dosing. This study is being done in people with normal kidney function and those with end-stage renal disease to see if they respond differently to the study drug.

DETAILED DESCRIPTION:
Specifically, the purpose of this study is to assess the influence of end-stage renal disease (ESRD) on area under the curve (both area under the curve, from time 0 to the last concentration measured [AUC0-last] and area under the curve, from time 0 extrapolated to infinity [AUC0-inf]) of carfilzomib 56 mg/m² at Cycle 2 Day 1 (C2D1) in patients with relapsed multiple myeloma.

ELIGIBILITY:
Key Inclusion Criteria:

1. Relapsed multiple myeloma
2. Evaluable disease (serum protein electrophoresis [SPEP]/urine protein electrophoresis [UPEP]/serum free light chain [SFLC] criteria)
3. Received at least 1 prior treatment regimen or line of therapy for multiple myeloma
4. End-stage renal disease (ESRD) on hemodialysis or CrCl ≥ 75 mL/min
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
6. Adequate organ and bone marrow function
7. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention or myocardial infarction within the protocol-specified period prior to enrollment

Key Exclusion Criteria:

1. Immunoglobulin M (IgM) multiple myeloma
2. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
3. Waldenström Macroglobulinemia
4. Active congestive heart failure (NYHA Class III-IV) ischemia, conduction abnormalities
5. Known human immunodeficiency virus (HIV), recent hepatitis B virus (HBV), hepatitis C virus (HCV)
6. Myelodysplastic Syndrome
7. Contraindication to test article, constituents, or required concomitant medications
8. Other investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (13):
- United States (6):
  - Karmanos Cancer Institute, Detroit, Michigan
  - North Shore-LIJ Health System/Center for Advanced Medicine - North Shore University Hospital, Lake Success, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Vanderbilt-Ingram Cancer Center, Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Malignant Haematology and Stem Cell Transplant Department, Melbourne, Victoria
- Canada (2):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Sir Mortimer B. Davis-Jewish General Hospital, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 13 investigative study centers (6 in the United States, 2 in Canada, and 5 in Australia) from 29 January 2014 to 25 March 2015.
  This study is ongoing, results are reported as of the data cut-off date of 12 October 2015.
Pre-assignment Details: Participants with relapsed multiple myeloma were enrolled into cohorts according to renal function (normal creatinine clearance (CrCl) or end-stage renal disease (ESRD; patients on hemodialysis)). Renal function was based on calculated CrCl using the Cockcroft-Gault formula at baseline.
Period: Overall Study
Arm/Group | Normal Renal Function | End Stage Renal Disease
Started | 15 | 11
Completed | 12 | 8
Not Completed | 3 | 3
Not completed — On-study at the Data Cut-off Date | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Normal Renal Function: Participants with normal renal function received carfilzomib 20 mg/m² IV on days 1 and 2 of cycle 1, followed by 27 mg/m² IV on days 8, 9, 15, and 16 of cycle 1. Participants who adequately tolerated dosing at 27 mg/m² received carfilzomib 56 mg/m² IV on days 1, 2, 8, 9, 15 and 16 of cycle 2 and all subsequent cycles.
- End Stage Renal Disease: Participants with ESRD received carfilzomib 20 mg/m² IV on days 1 and 2 of cycle 1, followed by 27 mg/m² IV on days 8, 9, 15, and 16 of cycle 1. Participants who adequately tolerated dosing at 27 mg/m² received carfilzomib 56 mg/m² IV on days 1, 2, 8, 9, 15 and 16 of cycle 2 and all subsequent cycles.
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | End Stage Renal Disease | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (8.1) | 62.8 (7.9) | 64.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 9 | 23
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 0 | 1
  Black | 1 | 1 | 2
  White | 12 | 9 | 21
  Other | 1 | 0 | 1
  Not Reported | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active; 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, no self-care, confined to bed or chair; 5 = Dead.
  participants
    0 (Fully active) | 5 | 3 | 8
    1 (Restrictive but ambulatory) | 10 | 7 | 17
    2 (Ambulatory but unable to work) | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve From Time 0 to Last Concentration (AUC0-last) of Carfilzomib Following 56 mg/m² Carfilzomib on Day 1 of Cycle 2
Description: Carfilzomib plasma concentrations for pharmacokinetic (PK) analyses were measured by liquid chromatography with tandem mass spectrometry. The lower limit of quantitation (LLOQ) for the assay was 0.3 ng/mL.
Time Frame: Cycle 2, day 1 at predose, 15 minutes post start of infusion, immediately before the end of infusion, and at 5, 15, and 30 minutes, and 1, 2, and 4 hours after the end of the infusion.
Population: PK evaluable population for cycle 2, day 1. The PK evaluable population is defined as participants with sufficient carfilzomib plasma concentration versus time data for the estimation of PK parameters by non-compartmental analysis on cycle 1, day 16 and/or cycle 2, day 1. One participant was excluded due to samples taken from the infusion arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 10 | 8
ng*h/mL | 563 (41.9) | 747 (143.9)
Statistical Analysis 1: Comparison: Normal Renal Function vs End Stage Renal Disease; Test type: Superiority or Other; Ratio of geometric means = 132.75, 90% CI 2-sided [70.60 to 249.63] — The point estimates of the geometric mean ratios for the PK parameters were calculated by exponentiation of the differences in the least-squares means between the renal impairment group (test) and participants with normal renal function (reference)

2. Primary Outcome: Area Under the Concentration Time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of Carfilzomib Following 56 mg/m² Carfilzomib on Day 1 of Cycle 2
Time Frame: as for outcome 1
Population: PK evaluable population for cycle 2, day 1. One participant was excluded due to samples taken from the infusion arm, distal to the infusion site.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 10 | 8
ng*h/mL | 563 (41.8) | 752 (144.7)
Statistical Analysis 1: Comparison: Normal Renal Function vs End Stage Renal Disease; Test type: Superiority or Other; Ratio of geometric means = 133.62, 90% CI 2-sided [70.93 to 251.73]

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Carfilzomib Following 56 mg/m² Carfilzomib on Day 1 of Cycle 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 10 | 8
ng/mL | 1389 (26.8) | 1567 (128.8)

4. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Carfilzomib Following 56 mg/m² Carfilzomib on Day 1 of Cycle 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 10 | 8
hours | 0.467 [0.250 to 0.733] | 0.467 [0.250 to 0.583]

5. Secondary Outcome: Terminal Half-life (T½) of Carfilzomib Following 56 mg/m² Carfilzomib on Day 1 of Cycle 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 10 | 8
hours | 0.341 [0.111 to 0.498] | 1.25 [0.0632 to 3.31]

6. Secondary Outcome: Clearance (CL) of Carfilzomib Following 56 mg/m² Carfilzomib on Day 1 of Cycle 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 10 | 8
liters/hour | 179 (38.9) | 134 (136.9)

7. Secondary Outcome: Mean Residence Time (MRT) of Carfilzomib Following 56 mg/m² Carfilzomib on Day 1 of Cycle 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 10 | 8
hours | 0.135 (62.6) | 0.245 (79.9)

8. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Carfilzomib Following 56 mg/m² Carfilzomib on Day 1 of Cycle 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 10 | 8
liters | 24.1 (44.8) | 32.8 (133.9)

9. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to Last Concentration (AUC0-last) of Carfilzomib Following 27 mg/m² Carfilzomib on Day 16 of Cycle 1
Time Frame: Cycle 1, day 16 at predose, 15 minutes post start of infusion, immediately before the end of infusion, and at 5, 15, and 30 minutes, and 1, 2, and 4 hours after the end of the infusion.
Population: PK evaluable population for cycle 1, day 16. One participant was excluded due to samples taken from the infusion arm, distal to the infusion site.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
ng*h/mL | 344 (24.8) | 480 (36.0)

10. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of Carfilzomib Following 27 mg/m² Carfilzomib on Day 16 of Cycle 1
Time Frame: as for outcome 9
Population: PK evaluable population for cycle 1, day 16. One participant was excluded due to samples taken from the infusion arm, distal to the infusion site. Participants for whom the coefficient of correlation (R²) was < 0.8 were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 11 | 6
ng*h/mL | 347 (26.3) | 479 (46.6)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Carfilzomib Following 27 mg/m² Carfilzomib on Day 16 of Cycle 1
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
ng/mL | 819 (29.8) | 1022 (37.2)

12. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Carfilzomib Following 27 mg/m² Carfilzomib on Day 16 of Cycle 1
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
hours | 0.583 [0.467 to 0.733] | 0.467 [0.233 to 0.750]

13. Secondary Outcome: Terminal Half-life (T½) of Carfilzomib Following 27 mg/m² Carfilzomib on Day 16 of Cycle 1
Time Frame: as for outcome 9
Population: PK evaluable population for cycle 1, day 16. One participant was excluded due to samples taken from the infusion arm, distal to the infusion site. Participants with a coefficient of correlation (R²) < 0.8 were excluded.
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 11 | 6
hours | 0.387 [0.0938 to 0.599] | 0.992 [0.918 to 16.0]

14. Secondary Outcome: Clearance (CL) of Carfilzomib Following 27 mg/m² Carfilzomib on Day 16 of Cycle 1
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
liters/hour | 146 (23.0) | 93 (56.8)

15. Secondary Outcome: Mean Residence Time (MRT) of Carfilzomib Following 27 mg/m² Carfilzomib on Day 16 of Cycle 1
Time Frame: as for outcome 9
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 11 | 6
hours | 0.222 (16.6) | 0.426 (152.2)

16. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Carfilzomib Following 27 mg/m² Carfilzomib on Day 16 of Cycle 1
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
liters | 32.0 (29.7) | 53.0 (185.5)

17. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to Last Concentration (AUC0-last) for Metabolite PR-389/M14
Time Frame: Cycle 1, day 16 and cycle 2, day 1 at predose, 15 minutes post start of infusion, immediately before the end of infusion, and at 5, 15, and 30 minutes, and 1, 2, and 4 hours after the end of the infusion.
Population: PK evaluable population; One participant was excluded due to samples taken from the infusion arm, distal to the infusion site. "n" indicates the number of participants included in the analyses at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
ng*h/mL
  Cycle 1, Day 16 (n = 13, 9) | 320 (32.8) | 1486 (32.3)
  Cycle 2, Day 1 (n = 10, 8) | 584 (17.5) | 2086 (132.8)

18. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) for Metabolite PR-389/M14
Time Frame: as for outcome 17
Population: PK evaluable population. Participants for whom the extrapolated portion of AUC0-∞ was > 20% were excluded. AUC0-∞ could not be calculated for the ESRD group as the extrapolated portion (AUCextr) was greater than 20% in all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 10 | 0
ng*h/mL
  Cycle 1, Day 16 | 355 (25.1) |
  Cycle 2, Day 1 | 650 (22.5) |

19. Secondary Outcome: Maximum Observed Plasma Concentration for Metabolite PR-389/M14
Time Frame: as for outcome 17
Population: PK evaluable population; one participant was excluded due to samples taken from the infusion arm, distal to the infusion site.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
ng/mL
  Cycle 1, Day 16 (n = 13, 9) | 153 (25.4) | 413 (32.9)
  Cycle 2, Day 1 (n = 10, 8) | 302 (16.5) | 595 (128.4)

20. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) for Metabolite PR-389/M14
Time Frame: as for outcome 17
Population: as for outcome 19
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
hours
  Cycle 1, Day 16 (n = 13, 9) | 1.00 [0.750 to 1.13] | 1.50 [1.00 to 2.67]
  Cycle 2, Day 1 (n = 10, 8) | 0.983 [0.583 to 1.02] | 2.00 [1.45 to 4.47]

21. Secondary Outcome: Terminal Half-life (T½) of Metabolite PR-389/M14
Time Frame: as for outcome 17
Population: PK evaluable population. Participants for whom the extrapolated portion of AUC0-∞ was > 20% were excluded. T½ could not be calculated for the ESRD group as the extrapolated portion (AUCextr) was greater than 20% in all participants.
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 10 | 0
hours
  Cycle 1, Day 16 | 1.46 [0.975 to 1.73] |
  Cycle 2, Day 1 | 1.10 [0.903 to 1.70] |

22. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to Last Concentration (AUC0-last) for Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
ng*h/mL
  Cycle 1, Day 16 (n = 13, 9) | 33.4 (53.9) | 54.6 (45.0)
  Cycle 2, Day 1 (n = 10, 8) | 60.3 (48.4) | 86.3 (199.1)

23. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) for Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: PK evaluable population. One participant was excluded due to samples taken from the infusion arm, distal to the infusion site. Participants for whom the extrapolated portion of AUC0-∞ was > 20% were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 7
ng*h/mL
  Cycle 1, Day 16 (n = 13, 7) | 36.2 (54.1) | 66.4 (48.7)
  Cycle 2, Day 1 (n = 10, 5) | 63.8 (48.0) | 131 (35.8)

24. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
ng/mL
  Cycle 1, Day 16 (n = 13, 9) | 20.7 (43.5) | 25.9 (42.5)
  Cycle 2, Day 1 (n = 10, 8) | 40.2 (38.5) | 42.3 (163.9)

25. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) for Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: as for outcome 19
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
hours
  Cycle 1, Day 16 (n = 13, 9) | 0.833 [0.683 to 1.00] | 0.767 [0.733 to 1.05]
  Cycle 2, Day 1 (n = 10, 8) | 0.667 [0.250 to 1.00] | 0.750 [0.717 to 1.52]

26. Secondary Outcome: Terminal Half-life (T½) of Metabolite PR-413/M15
Time Frame: as for outcome 17
Population: as for outcome 23
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 7
hours
  Cycle 1, Day 16 (n = 13, 7) | 1.07 [0.544 to 1.33] | 1.41 [1.30 to 1.86]
  Cycle 2, Day 1 (n = 10, 5) | 0.962 [0.802 to 1.21] | 1.37 [1.04 to 1.44]

27. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to Last Concentration (AUC0-last) for Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
ng*h/mL
  Cycle 1, Day 16 (n = 13, 9) | 82.8 (53.1) | 86.8 (44.3)
  Cycle 2, Day 1 (n = 10, 8) | 147 (52.8) | 138 (126.6)

28. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) for Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
ng*h/mL
  Cycle 1, Day 16 (n = 13, 9) | 84.4 (52.4) | 89.6 (42.8)
  Cycle 2, Day 1 (n = 10, 8) | 148 (51.7) | 139 (125.1)

29. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
ng/mL
  Cycle 1, Day 16 (n = 13, 9) | 93.4 (40.2) | 90.4 (48.0)
  Cycle 2, Day 1 (n = 10, 8) | 180 (40.5) | 151 (129.7)

30. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) for Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: as for outcome 19
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
hours
  Cycle 1, Day 16 (n = 13, 9) | 0.617 [0.467 to 1.00] | 0.600 [0.467 to 0.917]
  Cycle 2, Day 1 (n = 10, 8) | 0.525 [0.250 to 0.617] | 0.533 [0.467 to 0.750]

31. Secondary Outcome: Terminal Half-life (T½) of Metabolite PR-519/M16
Time Frame: as for outcome 17
Population: as for outcome 19
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 13 | 9
hours
  Cycle 1, Day 16 (n = 13, 9) | 0.705 [0.473 to 0.993] | 0.721 [0.518 to 1.42]
  Cycle 2, Day 1 (n = 10, 8) | 0.617 [0.555 to 0.673] | 0.687 [0.473 to 0.933]

32. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Determination of the severity of all adverse events was assessed following the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.03, where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Fatal.
  A Serious AE is an AE that meets one or more of the following criteria:
  * Death,
  * Life-threatening experience;
  * Requires in-patient hospitalization or prolongation of an existing hospitalization,
  * Results in persistent or significant disability/incapacity,
  * Is a congenital anomaly/birth defect,
  * Important medical events that may not result in death, be life-threatening, or require hospitalization.
  Treatment-related adverse events (TRAEs) are adverse events considered related to carfilzomib by the investigator, including those with unknown relationship.
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug as of the data cut-off date of 12 October 2015; median duration of treatment was 14 weeks in the normal renal function group and 12 weeks in the ESRD group.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | End Stage Renal Disease
Number analyzed (Participants) | 15 | 11
participants
  Any adverse event | 15 | 11
  Adverse event ≥ Grade 3 | 12 | 9
  Serious adverse event | 10 | 9
  AE leading to discontinuation of carfilzomib | 6 | 0
  Fatal adverse events | 2 | 1
  Treatment-related adverse events | 12 | 8
  Treatment-related adverse event ≥ Grade 3 | 7 | 6
  Serious treatment-related adverse event | 5 | 2
  TRAE leading to discontinuation of carfilzomib | 4 | 0
  Treatment-related fatal adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after the last dose of study drug as of the data cut-off date of 12 October 2015; median duration of treatment was 14 weeks in the normal renal function group and 12 weeks in the ESRD group.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Normal Renal Function | End Stage Renal Disease
Serious Adverse Events (participants affected / at risk) | 10/15 | 9/11
Other Adverse Events (participants affected / at risk) | 14/15 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=15) | End Stage Renal Disease (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Death (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 3 | 2
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Troponin increased (Investigations) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=15) | End Stage Renal Disease (N=11)
Anaemia (Blood and lymphatic system disorders) | 8 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1
Ear congestion (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Exophthalmos (Eye disorders) | 1 | 0
Eye discharge (Eye disorders) | 0 | 1
Eye inflammation (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Eye swelling (Eye disorders) | 2 | 0
Eyelid oedema (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0
Ocular discomfort (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 5
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mouth swelling (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 6
Retching (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4
Application site reaction (General disorders) | 1 | 0
Catheter site inflammation (General disorders) | 0 | 1
Chest discomfort (General disorders) | 2 | 1
Chest pain (General disorders) | 2 | 0
Chills (General disorders) | 3 | 1
Fatigue (General disorders) | 8 | 5
General physical health deterioration (General disorders) | 2 | 0
Influenza like illness (General disorders) | 1 | 0
Infusion site erythema (General disorders) | 1 | 0
Infusion site pain (General disorders) | 2 | 0
Injury associated with device (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 8 | 2
Sluggishness (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Respiratory tract infection (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 0 | 1
Blood calcium increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
Carbon dioxide decreased (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Monocyte count decreased (Investigations) | 0 | 1
Monocyte count increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Olfactory test abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Protein total decreased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Areflexia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 3
Lethargy (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 1
Mood altered (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 2 | 2
Peripheral coldness (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.